CLINICAL TRIAL: NCT00284661
Title: Meniscal Repair: A Randomized Prospective Trial of FAST-FIX vs. Meniscal Suturing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fowler Kennedy Sport Medicine Clinic (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11125; R3773A01 (Other Grant/Funding Number: Smith and Nephew)
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Meniscal Tear
Keywords: Meniscal repair; Meniscal suturing; Meniscal tear

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FAST FIX (Experimental): Inetrvention is Fast Fix repair of meniscal tear
  Interventions: Procedure: FAST FIX
- Meniscal suturing (Experimental): Intervention is Standard suturing of meniscal tear
  Interventions: Procedure: Meniscal suturing

INTERVENTIONS:
Procedure: FAST FIX — Fast fix repair of a meniscal tear
  Arms: FAST FIX
Procedure: Meniscal suturing — standard suturing of meniscal tear
  Arms: Meniscal suturing

SUMMARY:
Meniscal repair resulting in meniscal preservation is the most desirable treatment of a torn meniscus and is one of the most commonly performed arthroscopic procedures. The inside-out meniscal suturing technique allows precise placement of sutures under direct visualization and studies have reported excellent healing rates and low re-tear rates. However, complications associated with the use of the inside-out technique (injury to the knee's neurovascular structures and infection) and the fact that it is a time consuming procedure have generated the development of alternative methods and devices. The FasT-Fix is reported to be quicker and safer. It is applicable to tears in most locations and requires no additional incisions or portals. Even though this and many similar devices are widely used with reported clinical healing rates of 75 -92% and relatively minor complications, few prospective, randomized clinical trials evaluating and comparing different techniques have been carried out. Patient outcome studies are necessary to evaluate which technique ultimately results in the most effective repair and the least patient disability following surgery.

We hypothesize that an inside-out suturing technique will have a higher complication rate but a significantly lower failure rate than the FasT-Fix Menisical Repair System

DETAILED DESCRIPTION:
In this prospective, randomized, trial subjects will be randomly assigned to the inside-out group or the FasT-Fix group and will be followed for at least 24 months. Primary outcome is the difference between groups in the disease specific quality of life assessment - The Western Ontario Meniscal Evaluation Tool. Secondary outcome measures include range of motion, functional outcome scores, surgical time, complication rate, meniscal retear and differences between groups in post-operative pain. The data collector will be blinded to patients' intervention group. Secondary outcome measures include range of motion, functional outcome scores, disease-specific quality of life outcome scores and the standard knee clinical examination.

Study Population: The investigators will assess all patients presenting with suspected meniscal tears. Those meeting the inclusion/exclusion criteria will be asked to sign an informed consent. Subjects who have successfully been screened and are slated to be randomized into the study must have a pre-operative visit within 12 months of their scheduled surgery.

Routine knee x-rays will be performed on all patients to rule out extensive degenerative changes, loose bodies, fractures, osteochondritis dissecans and other lesions.

Treatment Protocols: Intervention group assignment will take place at the time of surgery, once the patient has undergone the initial arthroscopy and a diagnosis of a repairable meniscal tear has been confirmed. Patients will be stratified for surgeon and for concurrent ACL reconstruction. They will then be randomized to one of the two treatment groups.

Meniscal repair is a day surgery procedure performed under general anaesthesia and tourniquet control as required. Prior to the repair, synovial abrasion and debridement of scar tissue will be carried out to promote vascular ingrowth.

FasT-Fix Technique A suture that is pre-attached to a T-bar is placed across the meniscal tear via a sheathed needle. A small obturator pushes the "T" out of the needle engaging the outer rim of the meniscus in the synovial recess. The suture tails are tied arthroscopically, stabilizing the tear.

Inside-Out Suturing Technique Repairs of the medial meniscus will be carried out with the knee in 10-30° flexion. This allows both preservation of the posterior capsular recess and full knee extension once the repair is complete. A vertical incision is made posterior to the medial collateral ligament. The deep fascia is incised and the posteromedial capsule visualized. The lateral meniscus is repaired through a vertical incision posterior to the lateral collateral ligament made with the knee flexed 90°. The iliotibial band is split in line with its fibers at the level of the joint line. The biceps femoris and lateral gastrocnemius tendon are retracted posteriorly, protecting the common peroneal nerve and exposing the capsule and popliteus tendon. Vertical sutures will be placed in at 5mm intervals along the tear. Sutures are tied over the capsule once ligamentous reconstruction, if necessary, is completed. This is done with the knee in full extension.

Assessments: Patients will be assessed pre-operatively and by a blinded research assistant at 3, 6, 12, and 24 months. A tubi-grip will cover the operative knee in order that the data collector may be blinded to treatment group. Effusion and joint-line tenderness will be assessed by the physician prior to the data collector's appraisal. The viability of the meniscal repair will be based on the clinical examination. The absence of effusion, joint-line tenderness and locking all correlate well with a healed meniscus. The International Knee Documentation Form, the Western Ontario Meniscal Evaluation Tool and the Lysholm score, validated measures for knee problems will be utilized. Patients will be asked to complete a pain journal for a period of 2 weeks following their surgery.

ELIGIBILITY:
Inclusion Criteria:

-** Canadians Only can be recruited for this trial

* History indicative of meniscal pathology (i.e. pain, locking, clicking or giving way of the knee) +/- ACL insufficiency
* On physical exam, evidence of a meniscal tear (i.e. a locked joint, joint line tenderness and pain on meniscal compression +/- evidence of an ACL tear
* Vertical tears in the peripheral 0-5mm of the meniscus that are reducible

Exclusion Criteria:

* Intraarticular/Extraarticular knee infection
* Metabolic bone, collagen, crystalline joint or neoplastic disease
* Previous meniscal repair
* Meniscal tears that are in the avascular zone
* Stable meniscal tears, i.e. tears <10mm and displaced < 3mm, partial tears
* Radial, horizontal or flap tears
* Unwillingness to comply with the rehabilitation protocol or to be followed for 2 years
* Inability or unwillingness of subject /legal guardian to give written informed consent

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2005-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Quality of life at 2 years as measured by The Western Ontario Meniscal Evaluation Tool (WOMET) | 2 years

SECONDARY OUTCOMES:
Side-to-side difference in knee joint range of motion | 2 years
Other physical symptoms such as joint line pain/tenderness, knee effusion | 2 years
Re-tear rate (as confirmed by MRI or arthroscopy), Functional outcome scores | 2 years
Surgical time | day 0
Complication rate | 2 years
Differences between groups in post-operative pain | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Willits, MD, Principal Investigator — The University of Western Ontario
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, University of Western Ontario, London, Ontario, Canada